CLINICAL TRIAL: NCT01858506
Title: Development and Evaluation of Lifestyle Assessment and Educational Tools for Diabetic People With Limited Literacy
Brief Title: Diabetes Lifestyle Assessment and Educational Tools
Acronym: I-ACE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ofra Kalter-Leibovici MD (Other Government)
Collaborators: The Gertner Institute (Other); Clalit Health Services (Other); European Foundation for the Study of Diabetes (Other)
Responsible Party: Sponsor-Investigator, Ofra Kalter-Leibovici MD, Director of the Unit of Cardiovascular Epidemiology, The Gertner Institute for Epidemiology & Health Policy Research., Sheba Medical Center
Organization: Sheba Medical Center (Other Government)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EFSD_I-ACE; 8677-11-SMC (Other: Sheba Medical Center Helsinki Committee)
Record Dates: First submitted 2013-05-12; First posted 2013-05-21 (Estimated); Last update posted 2016-04-15 (Estimated); Status verified 2016-04

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Type 2 diabetes mellitus; Lifestyle counselling; Lifestyle assessment; Randomized controlled trial; Diabetes education
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- I-ACE intervention arm (Experimental): lifestyle counselling using the interactive assessment, counselling and education (I-ACE)-based method.
  Interventions: Procedure: I-ACE intervention
- Standard lifestyle advice arm (Active Comparator): lifestyle counselling using the standard lifestyle advice (SLA) program currently provided to Clalit Health Services patients.
  Interventions: Procedure: Standard Lifestyle Advice

INTERVENTIONS:
Procedure: I-ACE intervention — lifestyle counselling using the interactive assessment, counselling and education (I-ACE)-based method.
  Arms: I-ACE intervention arm
Procedure: Standard Lifestyle Advice — lifestyle counselling using the standard lifestyle advice (SLA) program currently provided to Clalit Health Services patients.
  Arms: Standard lifestyle advice arm

SUMMARY:
Aim: To evaluate a culturally-adapted method of lifestyle assessment, counseling, and education among Arab people with diabetes who have varying literacy skills using an interactive computerized tool and graphically-enhanced patient logs for dietary and physical activity.

The investigators hypothesize that this tool will: a) increase patients' knowledge and understanding of the role of lifestyle (diet and physical activity) in diabetes management; b) improve patients' engagement in monitoring dietary intake and physical activity; c) improve dietary and physical activity behaviors and self-blood glucose monitoring (SBGM) practices; d) improve glycemic control; and, e) improve the efficiency of lifestyle assessment, education and counseling while increasing patients' engagement in the process.

DETAILED DESCRIPTION:
Aim: To evaluate a culturally-adapted method of lifestyle assessment, counseling, and education among Arab people with diabetes who have varying literacy skills using an interactive computerized tool and graphically-enhanced patient logs for dietary and physical activity. The investigators will evaluate the effectiveness of this method for: a) increasing patients' knowledge and understanding of the role of lifestyle (diet and physical activity) in diabetes management; b) improving patients' engagement in monitoring dietary intake and physical activity; c) improving dietary and physical activity behaviors and self-blood glucose monitoring (SBGM) practices; d) improving glycaemic control; and, e) improving the efficiency of lifestyle assessment, education and counseling while increasing patients' engagement in the process.

ELIGIBILITY:
Inclusion Criteria:

* 40-64 years old
* BMI 27-45 kg/m2
* Diagnosis of type 2 diabetes mellitus in medical record
* HbA1c 8.0%-11.5%

Exclusion Criteria:

* Short-acting insulin treatment
* Inadequate control of co-morbid conditions
* Factors that may limit adherence to interventions (e.g., any medical or physical condition that limits the ability to participate in physical activity or standard diets recommended for people with diabetes, pregnancy, uncontrolled psychiatric condition, significant cognitive impairment, blindness).

Ages: 40 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2014-08; Primary Completion 2016-02 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Change in lifestyle knowledge | Baseline, 3rd,6th,12th months
  Change in diabetes-related lifestyle (diet and physical activity) knowledge, will be assessed with a diet knowledge questionnaire specially adapted for this population. Change in physical activity knowledge will be measured with the SKILLD diabetes knowledge questionnaire.

SECONDARY OUTCOMES:
Patients' lifestyle monitoring | 1st,2nd,3rd,6th months
  Patient engagement in monitoring diet intake and physical activity, assessed with 3-day dietary and physical activity records.
Dietary and physical activity behaviours | Baseline and 12 months.
  Dietary and physical activity behaviours, assessed with food frequency and physical activity questionnaires.
SBGM practices | 1st, 2nd, 3rd, 6th, 12th months.
  Self Blood Glucose Monitoring practices. Information will be downloaded from the blood glucose meters' memory.
Glycaemic control | Baseline, 3rd,6th, and 12th months.
  Glycaemic control, assessed with HbA1c levels.
Weight and waist circumference | Baseline, 3rd, 6th, and 12th months.
  Change of weight and waist circumference during follow-up.

OTHER OUTCOMES:
Medical regimen for diabetes management | Baseline, 1st, 2nd, 3rd, 6th, and 12th month.
  Medical regimen for diabetes management, i.e. self-reported medical treatment for diabetes.

CONTACTS AND LOCATIONS:
Overall Officials: Ofra Kalter-Leibovici, M.D., Principal Investigator — Sheba Medical Center, the Gertner Institute for Epidemiology & Health Policy Research; Kathleen Abu-Saad, Ph.D., Principal Investigator — Gertner Institute for Epidemiology & Health Policy Research
Locations (1):
- Clalit Health Services, Shomron administration, Hadera, Israel

REFERENCES:
- [Derived] Abu-Saad K, Murad H, Barid R, Olmer L, Ziv A, Younis-Zeidan N, Kaufman-Shriqui V, Gillon-Keren M, Rigler S, Berchenko Y, Kalter-Leibovici O. Development and Efficacy of an Electronic, Culturally Adapted Lifestyle Counseling Tool for Improving Diabetes-Related Dietary Knowledge: Randomized Controlled Trial Among Ethnic Minority Adults With Type 2 Diabetes Mellitus. J Med Internet Res. 2019 Oct 16;21(10):e13674. doi: 10.2196/13674. PMID 31621640